CLINICAL TRIAL: NCT00928512
Title: A 16-week Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose-finding Study to Evaluate the Efficacy, Safety and Tolerability of Subcutaneous Secukinumab (AIN457) Followed by an Extension Phase up to a Total of 60 Weeks in Patients With Active Rheumatoid Arthritis Despite Stable Treatment With Methotrexate
Brief Title: Efficacy, Safety and Tolerability of AIN457 in Patients With Rheumatoid Arthritis (RA) Taking Methotrexate (MTX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457F2201; 2009-011000-34 (EudraCT Number)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, RA, ACR, inflammatory joints
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Secukinumab 25mg (Experimental): Secukinumab 25mg s.c. q4wk
  Interventions: Drug: Secukinmab
- Secukinumab 75mg (Experimental): Secukinumab 75mg s.c. q4wk
  Interventions: Drug: Secukinmab
- Secukinumab 150mg (Experimental): Secukinumab 150mg s. c. q4wk
  Interventions: Drug: Secukinmab
- Secukinumab 300mg (Experimental): Secukinumab 300mg s.c. q4wk
  Interventions: Drug: Secukinmab
- Secukinumab Placebo (Placebo Comparator): Secukinumab Placebo s.c. q4wk
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinmab — Secukinumab was supplied as a 150mg lyophiized cake in individual glass vials each. The study drug dose levels were 25mg, 75mg, 150mg and 300mg and was administered subcutaneously.
  Other Names: AIN457
  Arms: Secukinumab 150mg; Secukinumab 25mg; Secukinumab 300mg; Secukinumab 75mg
Drug: Placebo — Secukinumab placebo was supplied as a 150mg lyophiized cake in individual glass vials each. The placebo dose levels were 25mg, 75mg, 150mg and 300mg and was administered subcutaneously.
  Arms: Secukinumab Placebo

SUMMARY:
This study will assess at Week 16 the efficacy and safety of AIN457 at different doses in patients with active RA despite stable MTX therapy. Treatment will continue up to Week 48 with a safety follow-up at Week 60 to assess the long term efficacy and safety of AIN457 treatment in combination with MTX in RA.

ELIGIBILITY:
Inclusion Criteria:

* Presence of RA classified by ACR 1987 revised criteria. Patients with active RA should have been on MTX for at least 3 months and must currently be treated with a stable dose of MTX (> or =7.5 mg/week - < or = 25 mg/week) for at least 4 weeks
* At Baseline: Disease activity criteria defined by > or = 6 out of 28 tender joints and > or = 6 out of 28 swollen joints WITH either Screening value of hsCRP > or = 10 mg/L OR ESR > or = 28 mm/1st hr

Exclusion Criteria:

* RA patients functional status class IV classified according to the ACR 1991 revised criteria
* Patients taking high potency opioid analgesics (e.g., methadone, hydromorphone, or morphine)
* Any therapy by intra-articular injections (e.g. corticosteroid) required for treatment of acute RA flare within 4 weeks before randomization

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (13):
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
- Novartis Investigative Site, Brussels, Belgium
- Czechia (4):
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Prague
- Germany (5):
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, München
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Gyula
- Japan (5):
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Kawagoe, Saitama
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lublin
- Russia (5):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Yaroslavl
- Slovakia (3):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Piešťany, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
- South Korea (4):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (5):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City

REFERENCES:
- [Derived] Genovese MC, Durez P, Richards HB, Supronik J, Dokoupilova E, Aelion JA, Lee SH, Codding CE, Kellner H, Ikawa T, Hugot S, Ligozio G, Mpofu S. One-year efficacy and safety results of secukinumab in patients with rheumatoid arthritis: phase II, dose-finding, double-blind, randomized, placebo-controlled study. J Rheumatol. 2014 Mar;41(3):414-21. doi: 10.3899/jrheum.130637. Epub 2014 Jan 15. PMID 24429175
- [Derived] Genovese MC, Durez P, Richards HB, Supronik J, Dokoupilova E, Mazurov V, Aelion JA, Lee SH, Codding CE, Kellner H, Ikawa T, Hugot S, Mpofu S. Efficacy and safety of secukinumab in patients with rheumatoid arthritis: a phase II, dose-finding, double-blind, randomised, placebo controlled study. Ann Rheum Dis. 2013 Jun;72(6):863-9. doi: 10.1136/annrheumdis-2012-201601. Epub 2012 Jun 23. PMID 22730366

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 patients discontinued prior to Week 16.At Week 20, all patients on secukinumab 25-150 mg who were responders continued on their randomized dose regimens. Non-responders in the 25 mg and 75 mg groups were up-titrated to 150 mg and non-responders in the 150 mg group were up-titrated to 300 mg.
Groups:
- Secukinumab 150mg: Secukinumab 150mg s.c. q4wk
Period: Overall Study
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Started | 41 | 43 | 49 | 54 | 50
Discontinued Prior to Week 16 | 3 | 0 | 2 | 6 | 5
Reassigned at Week 20 (Non-responders) | 0 (All patients in the 300 mg group at Week 20 remained at this dose in this group.) | 23 (Non-responders in the AIN457 150 mg group were reassigned treatment to the 300 mg group.) | 23 (Non-responders in the AIN457 75 mg group were reassigned treatment to the 150 mg group.) | 27 (Non-responders in the AIN457 25 mg group were reassigned treatment to the 150 mg group.) | 45 (All placebo patients (responders & non-responders) were reassigned treatment to the 150 mg group.)
Not Reassigned at Week 20 (Responders) | 37 | 20 | 23 | 18 | 0
New Groups After Reassignment | 60 (1 patient in this group continued at Week 16 but did not receive any study drug at Week 20.) | 115 | 23 (1 patient in this group continued at Week 16 but did not receive any study drug at Week 20.) | 18 (2 patients in this group continued at Week 16 but did not receive any study drug at Week 20) | 0
Completed Week 16 | 38 | 43 | 47 | 48 | 45
Entered/Continued to Week 20 (All) | 37 | 43 | 46 | 45 | 45
Completed | 31 | 37 | 38 | 33 | 35
Not Completed | 10 | 6 | 11 | 21 | 15
Not completed — Adverse Event | 4 | 3 | 2 | 8 | 6
Not completed — Lack of Efficacy | 2 | 0 | 4 | 7 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 4 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1 | 3
Not completed — Administrative Problems | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set was defined as all subjects being randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo | Total
Number analyzed (Participants) | 41 | 43 | 49 | 54 | 50 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.61) | 57.8 (11.23) | 54.3 (9.84) | 53.3 (11.44) | 55.0 (10.46) | 54.9 (10.75)
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0
  >=18 - < 41 years | 3 | 3 | 4 | 6 | 6 | 22
  >=41 - < 65 years | 30 | 27 | 37 | 41 | 34 | 169
  >=65 - < 75 years | 7 | 11 | 8 | 6 | 9 | 41
  >=75 years | 1 | 2 | 0 | 1 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 38 | 45 | 34 | 183
  Male | 10 | 8 | 11 | 9 | 16 | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 32 | 30 | 37 | 38 | 39 | 176
  Black | 0 | 0 | 1 | 1 | 1 | 3
  Asian | 8 | 11 | 9 | 14 | 8 | 50
  Native American | 0 | 0 | 1 | 0 | 0 | 1
  Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 1 | 1 | 2 | 7
Geographical Region [Number; unit: Participants]
  East Asia | 8 | 11 | 9 | 13 | 8 | 49
  Non-East Asia | 33 | 32 | 40 | 41 | 42 | 188
Functional Status [Number; unit: Participants] — ACR classification criteria of functional status in rheumatoid arthritis: Class l: completely able to perform usual activities of daily living (self-care, vocational & avocational); Class ll: able to perform usual self-care and vocational activities but limited in avocational activities; Class lll: able to perform usual self-care activities but limited in vocational and avocational activities; Class IV: limited ability to perform usual self-care, vocational and avocational activities.
  Participants
    Class l | 2 | 3 | 2 | 5 | 4 | 16
    Class ll | 28 | 27 | 31 | 37 | 34 | 157
    Class lll | 11 | 13 | 16 | 12 | 12 | 64
    Class IV | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 78.9 (23.91) | 72.1 (16.52) | 74.3 (15.70) | 71.3 (14.16) | 75.9 (15.61) | 74.3 (17.27)
Weight Group [Number; unit: Participants]
  <90 kg | 32 | 35 | 40 | 50 | 40 | 197
  >=90 kg | 9 | 8 | 9 | 4 | 10 | 40
Height [Mean (Standard Deviation); unit: cm] | 163.3 (10.03) | 161.9 (10.84) | 165.4 (9.52) | 163.2 (7.07) | 166.1 (7.62) | 164.0 (9.06)
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 29.48 (8.383) | 27.32 (4.673) | 27.03 (4.936) | 26.69 (4.768) | 24.47 (5.229) | 27.52 (5.693)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology Response of 20 (ACR20) at 16 Weeks
Description: A participant was considered to have achieved the incidence of response (ACR20 criteria) if he/she had at least a 20% improvement in both the tender and swollen 28-joint counts and had at least 20% improvement in at least 3 of the following 5 measures: patient's assessment of rheumatoid athritis (RA) pain, patient's global assessment of disease activity, physician's global assessment of disease activity, patient's self-assesseddisability (Health Assessment Questionnaire [HAQ©] score)and acute phase rectant (C-reactive protein [hsCRP]/ESR).
Time Frame: 16cweeks
Population: Full analysis set (FAS) all subjects to whom study drug was assigned. Following the intent-to-treat principle, subjects were analyzed according to the treatment they were assigned to at randomization. FAS did not include subjects who have missing values for all post-baseline (visit >=3) assessments on all of the specified efficacy variables.
Measure: Number; unit: Participants
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
Participants | 22 | 20 | 23 | 18 | 18

2. Secondary Outcome: Number of Participants Who Achieved an ACR50 or ACR70 Response at Week 16
Description: A participant was considered as improved according to the ACR50 or ACR70 criteria if he/she had at least a 50% or 70% improvement, respectively, in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures: patient's assessment of rheumatoid athritis (RA) pain, patient's global assessment of disease activity, physician's global assessment of disease activity, patient self-assessed disability (Health Assessment Questionnaire [HAQ©] score) and Acute phase reactant (C-reactive protein [hsCRP]/ESR). Participants were defined as ACR50/70 responders at a given post-randomization visit if they satisfied the ACR50/70 criteria, respectively. Participants were considered ACR50/70 nonresponders if they failed the ACR50/70 criteria respectively. Participants who prematurely discontinued from study due to insufficient therapeutic effect were also considered nonresponders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
Participants
  ACR50 response | 7 | 9 | 9 | 8 | 3
  ACR70 response | 2 | 2 | 1 | 4 | 0

3. Secondary Outcome: Number of Participants Who Achieved an ACR20, ACR50 or ACR70 Response up to Week 16
Description: A participant was considered as improved according to the ACR20, ACR50 or ACR70 criteria if he/she had as least a 20%, 50% or 70% improvement, respectively, in both the tender and the swollen 28-joint count, and in at least 3 of the following 5 measures: patient's assessment of rheumatoid athritis (RA) pain, patient's global assessment of disease activity, physician's global assessment of disease activity, patient's self-assessed disability and acute phase rectant or Erythrocyte sedimentation rate (ESR).
Time Frame: at Weeks2, 4, 8, 12, 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
Participants
  Week 2: ACR20 response | 7 | 9 | 9 | 9 | 3
  Week 2: ACR50 response | 0 | 2 | 2 | 2 | 1
  Week 2: ACR70 response | 0 | 0 | 0 | 0 | 0
  Week 4: ACR20 response | 7 | 13 | 12 | 13 | 8
  Week 4: ACR50 response | 0 | 1 | 2 | 2 | 2
  Week 4: ACR70 response | 0 | 1 | 1 | 1 | 0
  Week 8: ACR20 response | 16 | 17 | 22 | 15 | 11
  Week 8: ACR50 response | 3 | 5 | 6 | 6 | 1
  Week 8: ACR70 response | 1 | 1 | 2 | 2 | 0
  Week 12: ACR20 response | 20 | 24 | 25 | 17 | 12
  Week 12: ACR50 response | 6 | 7 | 8 | 4 | 1
  Week 12: ACR70 response | 1 | 2 | 2 | 3 | 0
  Week 16: ACR20 response | 22 | 20 | 23 | 18 | 18
  Week 16: ACR50 response | 7 | 9 | 9 | 8 | 3
  Week 16: ACR70 response | 2 | 2 | 1 | 4 | 0

4. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Using CRP (DAS28-CRP)
Description: The DAS28 is a measure of disease activity in Rheumatoid Arthritis (RA). The score is calculated by a complex mathematical formula, which includes the number of tender and swollen joints (out of a total of 28), the erythrocyte sedimentation rate (ESR) or hsCRP, and the patient's 'global assessment of global health (indicated by marking a 100 mm line between very good and very bad). A DAS28 score greater than 5.1 implies active disease, less than 3.2 well controlled disease, and less than 2.6 remission. The DAS28-CRP was derived from swollen joint count, tender joint count, hsCRP and patient's global assessment of disease activity.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
scores on a scale | -1.29 (0.186) | -1.35 (0.181) | -1.46 (0.170) | -1.13 (0.165) | -0.96 (0.171)

5. Secondary Outcome: Change From Baseline in Medical Outcome Short Form (36) Health Survey (SF-36® v2)
Description: The SF-36 Scale is a 36-item, patient-reported survey which measures overall quality of life. It consists of 8 subscales (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health) which can be aggregated to derive a physical-component summary score and a mental-component score. Scores are normally determined with the use of norm-based methods which standardize scores based on an assessment of the general U.S. population free of chronic conditions. The scores range for each subscale from 0 to 10, and the composite score ranges from 0 to 100, with the higher scores indicative of better health.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale-change from baseline
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 48 | 52 | 47
scores on a scale-change from baseline
  SF-36 physical component score | 3.42 (5.574) [-2.66 to 3.60] | 4.51 (6.800) [-2.07 to 3.58] | 3.48 (5.961) [-2.05 to 3.32] | 2.15 (7.176) [-3.40 to 2.33] | 2.47 (7.481) [0.00 to 0.00]
  SF-36 mental component score | -0.76 (11.421) [-5.95 to 3.82] | 3.59 (9.631) [-3.08 to 4.41] | 2.58 (11.479) [-4.72 to 3.05] | 1.06 (9.299) [-2.07 to 5.03] | 1.10 (10.231) [0.00 to 0.00]

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at Week 16
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue©) is a 13- item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants responded to each item on a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much) based on their experience of fatigue during the past 2 weeThe scale score was computed by summing the item scores, after reversing those items that were worded in the negative direction. When there were missing item scores, the subscale score was computed by summing the non-missing item scores, multiplying by 13 (the total number of items in the scale) and dividing by the number of non-missing items. The latter rule applied only when at least half of the items (seven or more) were non-missing. FACIT-Fatigue subscale scores range from 0 to 52, where higher scores represent less fatigue.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale-change from baseline
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 48
scores on a scale-change from baseline | 2.80 (7.181) [-1.25 to 6.00] | 5.18 (8.470) [-2.00 to 5.00] | 3.89 (8.368) [-2.00 to 5.00] | 1.95 (8.232) [3.00 to 4.00] | 1.64 (8.464) [0.00 to 0.00]

7. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Week 16
Description: The distribution of EULAR response criteria was according to DAS28-CRP at Week 16. EULAR response criteria are based on DAS28-CRP status in combination with DAS28-CRP improvements. The EULAR response criteria are as follows: Week 16 DAS28-CRP <3.2 with DAS28-CRP improvement >1.2 corresponds to 'good response'; Week 16 DAS28-CRP <3.2 with DAS28-CRP improvement between 0.6 to 1.2, or Week 16 DAS28-CRP between 3.2 to 5.1 with DAS28-CRP improvement >1.2 or from 0.6 to 1.2, or WeeK 16 DAS28-CRP >5.1 with DAS28-CRP improvement >1.2 correspond to 'moderate response; Week 16 DAS28-CRP <3.2 with DAS28-CRP improvement <0.6, or Week 16 DAS28-CRP between 3.2 to 5.1 with DAS28-CRP improvement <0.6, or Week 16 DAS28-CRP >5.1 with DAS28-CRP improvement between 0.6 to 1.2 or <0.6 correspond to 'no response'.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
Percentage of participants
  Good Response | 19.5 | 18.6 | 22.4 | 18.9 | 14.3
  Moderate Response | 43.9 | 41.9 | 46.9 | 30.2 | 40.8
  No Response | 36.6 | 39.5 | 30.6 | 50.9 | 44.9

8. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF) Concentrations at Week 16
Description: Only values that were above normal range (12 U/mL) were were included.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 29 | 27 | 34 | 36 | 32
U/mL | -5.66 (210.235) | -32.11 (196.574) | -77.62 (341.985) | 66.44 (379.723) | 85.63 (499.964)

9. Secondary Outcome: Anti-CCP (Cyclic Citrulinated Peptide) Antibodies Concentrations at Baseline and at Week 16
Description: Only values that were above normal range (20 units) were included.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
Units
  Concentrations at baseline (n: 33, 32, 43, 46, 38) | 1444.67 (1450.438) | 1098.81 (1238.627) | 1178.88 (1390.458) | 1342.50 (1544.205) | 1406.79 (1496.032)
  Concentrations at Week 16 (n: 30, 30, 41, 42, 36) | 1478.53 (1767.070) | 1330.63 (1355.193) | 1155.27 (1550.003) | 1443.07 (1640.771) | 1556.06 (1596.122)

10. Secondary Outcome: Change From Baseline in ACR Component: Adjusted Swollen 28-joint Count at Week 16
Description: Synovial fluid and/or soft tissue swelling but not bony overgrowth represents a positive result for swollen joint count. Joint counts were performed according to the visit schedule by the physician or by well trained personnel. Whenever possible, the same evaluator performed these assessments at all visits. The following 28 joints were assessed for tenderness and swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). If the number of joints for which data were available (e.g., S) was less than 28, the number of swollen joints (e.g., s) was scaled up proportionately (i.e., 28*(s/S)).
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
swollen joints | -5.4 (0.75) | -5.2 (0.73) | -6.0 (0.68) | -4.4 (0.66) | -4.6 (0.69)

11. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Using ESR (DAS28-ESR) at Week 16
Description: The DAS28 is a measure of disease activity in Rheumatoid Arthritis (RA). The score is calculated by a complex mathematical formula, which includes the number of tender and swollen joints (out of a total of 28), the erythrocyte sedimentation rate (ESR) or hsCRP, and the patient's 'global assessment of global health (indicated by marking a 100 mm line between very good and very bad). A DAS28 score greater than 5.1 implies active disease, less than 3.2 well controlled disease, and less than 2.6 remission.The DAS28 was also derived using erythrocyte sedimentation rate (ESR) (referred to as DAS28-ESR).
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
scores on a scale | -1.48 (0.196) | -1.55 (0.191) | -1.65 (0.179) | -1.28 (0.174) | -1.14 (0.181)

12. Secondary Outcome: Change From Baseline in ACR Component: Adjusted Tender 28-joint Count at Week 16
Description: The ACR tender joint count (28 joints) was done by scoring several different aspects of tenderness as assessed by pressure and joint manipulation on physical examination. Joint counts were performed according to the visit schedule by the physician or by well trained personnel. The following 28 joints were assessed for tenderness and swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). If the number of joints for which data were available (e.g., T) was less than 28, the number of tender joints (e.g., t) was scaled up proportionately (i.e., 28*(t/T)).
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
tender joints | -6.3 (0.94) | -6.5 (0.91) | -6.3 (0.86) | -5.6 (0.83) | -5.0 (0.85)

13. Secondary Outcome: Change From Baseline in ACR Component: Patient's Assessment of RA Pain at Week 16
Description: The patient's assessment of pain was performed at all visits using 100 mm visual analog scale (VAS) ranging from "no pain" to "unbearable pain" after the question "Please indicate with a vertical mark ( | ) through the horizontal line the most pain you had from your rheumatoid arthritis over the last 24 hours.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: VAS in mm
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
VAS in mm | -9.0 (3.25) | -9.1 (3.16) | -11.6 (2.97) | -9.5 (2.88) | -9.1 (2.99)

14. Secondary Outcome: Change From Baseline in ACR Component: Patient's Global Assessment of Disease Activity at Week 16
Description: The patient's global assessment of disease activity was performed at the visits on a 100 mm non-anchored visual analog scale, from no arthritis (0) activity to maximal arthritis (100) activity, after the question, "Considering all the ways your arthritis affects you, draw a line on the scale for how well you are doing".
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: VAS in mm
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
VAS in mm | -10.1 (3.27) | -10.5 (3.19) | -18.4 (2.99) | -10.6 (2.90) | -9.9 (3.01)

15. Secondary Outcome: Change From Baseline in ACR Component: Physician's Global Assessment of Disease Activity at Week 16
Description: The physician's global assessment of disease activity was performed at the visits usingon a 100 mm non-anchored visual analog scale, from no arthritis (0) activity to maximal arthritis (100) activity, after the question, "Considering all the ways your arthritis affects you, draw a line on the scale for how well you are doing".
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: VAS in mm
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
VAS in mm | -22.8 (2.99) | -26.7 (2.91) | -25.4 (2.73) | -18.1 (2.65) | -15.2 (2.74)

16. Secondary Outcome: Change From Baseline in ACR Component: Health Assessment Questionnaire (HAQ©) Score at Week 16
Description: HAQ© was used to assess physical ability and functional status of patients as well as quality of life at the visits in these 8 categories assessed by the Disability Index: dressing & grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Patients report amount of difficulty they have in performing 2 or 3 specific activities. There are 4 possible responses (0, 1, 2, 3) for these questions which include types of assistance, if any; the participant uses for his/her usual activities: 0: without any difficulty- No assistance is needed; 1: with some difficulty - A special device is used by the patient in his/her usual activities; 2: with much difficulty - The patient usually needs help from another person. 3: Unable to do - the patient usually needs both a special device and help from another person. Scores of 0 - 1 are generally considered to represent mild to moderate difficulty, 1-2 moderate to severe disability, and 2 -3 severe to very severe disability.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
scores on a scale | -0.297 (0.0698) | -0.256 (0.0688) | -0.233 (0.0639) | -0.202 (0.0627) | -0.116 (0.0652)

17. Secondary Outcome: Change From Baseline in ACR Component: High Sensitivity C-reactive Protein (hsCRP)
Description: Blood for this assessment was obtained at the visits in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.Since the results of this test may have unblinded study personnel, results from the central lab were provided for screening and baseline only. The hsCRP results from samples collected during the treatment period were revealed only after final database lock.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
mg/L | -6.54 (2.237) | -7.76 (2.175) | -9.09 (2.042) | -4.08 (1.984) | 0.30 (2.035)

18. Secondary Outcome: Change From Baseline in ACR Component: Erythrocyte Sedimentation Rate (ESR) at Week 16
Description: Blood for ESR, which is helpful to diagnose inflammatory diseases and to monitor disease activity and response to therapy, was obtained at the visits.
Time Frame: Baseline, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm/hr
Arm/Group | Secukinumab 300mg | Secukinumab 150mg | Secukinumab 75mg | Secukinumab 25mg | Secukinumab Placebo
Number analyzed (Participants) | 41 | 43 | 49 | 53 | 50
mm/hr | -13.51 (2.630) | -15.06 (2.564) | -15.43 (2.426) | -9.86 (2.331) | -6.12 (2.395)

ADVERSE EVENTS:
Groups:
- AIN457 25mg: Up to Week 20 - AIN457 25mg
- AIN457 75mg: Up to Week 20 - AIN457 75mg
- AIN457 150mg: Up to Week 20 - AIN457 150mg
- AIN457 300mg: Up to Week 20 - AIN457 300mg
- Placebo: Up to Week 20 - Placebo
- AIN457 25mg (Wk 20 to End of Study): From week 20 through end of study - AIN457 25mg
- AIN457 75mg (Wk 20 to End of Study): From week 20 through end of study - AIN457 75mg
- AIN457 150mg (Wk 20 to End of Study): From week 20 through end of study - AIN457 150mg
- AIN457 300mg (Wk 20 to End of Study): From week 20 through end of study - AIN457 300mg
Arm/Group | AIN457 25mg | AIN457 75mg | AIN457 150mg | AIN457 300mg | Placebo | AIN457 25mg (Wk 20 to End of Study) | AIN457 75mg (Wk 20 to End of Study) | AIN457 150mg (Wk 20 to End of Study) | AIN457 300mg (Wk 20 to End of Study)
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/49 | 0/43 | 4/41 | 1/50 | 1/18 | 3/23 | 9/115 | 8/60
Other Adverse Events (participants affected / at risk) | 14/54 | 21/49 | 15/43 | 15/41 | 24/50 | 11/18 | 15/23 | 52/115 | 27/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 25mg (N=54) | AIN457 75mg (N=49) | AIN457 150mg (N=43) | AIN457 300mg (N=41) | Placebo (N=50) | AIN457 25mg (Wk 20 to End of Study) (N=18) | AIN457 75mg (Wk 20 to End of Study) (N=23) | AIN457 150mg (Wk 20 to End of Study) (N=115) | AIN457 300mg (Wk 20 to End of Study) (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 25mg (N=54) | AIN457 75mg (N=49) | AIN457 150mg (N=43) | AIN457 300mg (N=41) | Placebo (N=50) | AIN457 25mg (Wk 20 to End of Study) (N=18) | AIN457 75mg (Wk 20 to End of Study) (N=23) | AIN457 150mg (Wk 20 to End of Study) (N=115) | AIN457 300mg (Wk 20 to End of Study) (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 4 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 4 | 4 | 3 | 1 | 4 | 15 | 8
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 5
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 6 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 5 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Monocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0 | 2 | 2 | 0 | 6 | 3
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 3 | 1
Varicose ulceration (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.